CLINICAL TRIAL: NCT05860777
Title: Harnessing Health Information Technology to Promote Equitable Care for Patients with Limited English Proficiency and Complex Care Needs
Brief Title: Harnessing Health IT to Promote Equitable Care for Patients with Limited English Proficiency and Complex Care Needs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian W. Pickering, M.B., B.Ch., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-002926
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Artificial Intelligence
Keywords: Limited English Proficiency; Machine Learning; Language Barrier; Complex Medical Needs

STUDY DESIGN:
Intervention Model Description: This is a pragmatic clinical trial-a stepped wedge cluster randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This is the control group who receive standard of care
- Intervention (Experimental): This is the group in units who are identified via AI model and in which interpreter services are actively reaching out to clinicians
  Interventions: Other: Complexity score and implementation

INTERVENTIONS:
Other: Complexity score and implementation — AI machine learning model to identify patients with complex care needs and implementation with active reaching out to clinicians to offer interpreter services
  Other Names: AI machine learning model and implementation with reaching out to clinicians
  Arms: Intervention

SUMMARY:
This is a pragmatic trial that will measure if the use of AI to identify patients with complex care needs and language barriers, as well as active reaching out to clinicians to offer the use of interpreter services will improve the frequency of interpreter use and reduce the time to first interpreter use

ELIGIBILITY:
Inclusion Criteria:

* Adults with limited English proficiency and requiring an interpreter and having complex medical care needs (includes admitted to the ICU, prolonged hospital stay, requiring palliative care)
* Have research authorization

Exclusion Criteria:

- Do not require an interpreter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1923 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Number of interpreters | 12 months
  the number of interpreters used among patients with LEP and complex care needs

SECONDARY OUTCOMES:
Change in time to interpreter use | 12 months
  The time measured in hours and minutes for an interpreter to be used for patients with LEP

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pickering, MB, B.Ch, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barwise A, Strechen I, Eltalhi T, Piche K, Wilson P, Tschida-Reuter D, Liu E, Herasevich S, Schulte PJ, Sutor B, Pickering B. Improving In-person Interpreter Utilization in Complex Care: Findings from a Stepped-Wedge Cluster Randomized Trial of Integrated Artificial Intelligence. J Gen Intern Med. 2026 Jan 5. doi: 10.1007/s11606-025-10104-9. Online ahead of print. PMID 41491380
- [Derived] Strechen I, Wilson P, Eltalhi T, Piche K, Tschida-Reuter D, Howard D, Sutor B, Tiong I, Herasevich S, Pickering B, Barwise A. Harnessing health information technology to promote equitable care for patients with limited English proficiency and complex care needs. Trials. 2024 Jul 4;25(1):450. doi: 10.1186/s13063-024-08254-y. PMID 38961501
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials